CLINICAL TRIAL: NCT07203924
Title: Prognostic Importance of Physical Activity Level in Geriatric Patients With Acute Coronary Syndrome
Brief Title: Prognostic Importance of Physical Activity in Geriatric Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Özkan Işık, Professor, Balikesir University
Other Study IDs: 2024/192 (BU Ethics No)
Record Dates: First submitted 2025-09-12; First posted 2025-10-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndromes; Geriatric Patients; Physical Activity Levels
Keywords: Acute Coronary Syndrome; TIMI; HEART; SVEAT; Physical Activity
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric ACS Patients: This cohort consists of 207 patients aged 65 years and older who presented to the emergency department with acute coronary syndrome (ACS). No intervention was performed. Physical activity levels were assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF), and outcomes were compared with major adverse cardiac events (MACE), mortality, and risk scores (TIMI, HEART, SVEAT).

SUMMARY:
This observational study evaluated the relationship between physical activity level and prognosis in geriatric patients admitted to the emergency department with acute coronary syndrome (ACS). A total of 207 patients aged 65 years and older were included. Physical activity level was assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF) and compared with clinical outcomes and risk scores (TIMI, HEART, SVEAT). Results showed that patients with higher physical activity levels had lower rates of major adverse cardiac events (MACE) and mortality, as well as lower risk scores. The findings suggest that physical activity is an independent protective factor that improves prognosis in older patients with ACS.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) in elderly patients is associated with high morbidity and mortality, and identifying prognostic factors is clinically important. Physical activity is known to have protective cardiovascular effects, but its prognostic role in geriatric ACS patients remains unclear.

This observational study will include 207 patients aged 65 years and older who present to the emergency department with ACS. Physical activity levels will be measured using the International Physical Activity Questionnaire-Short Form (IPAQ-SF). Activity scores will then be compared with clinical outcomes, including major adverse cardiac events (MACE), mortality, and risk stratification scores (TIMI, HEART, SVEAT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Admission to the emergency department with a diagnosis of acute coronary syndrome (ACS)
* Ability to complete the International Physical Activity Questionnaire-Short Form (IPAQ-SF)

Exclusion Criteria:

* Age < 65 years
* Patients without ACS diagnosis
* Patients unable to complete the IPAQ-SF questionnaire (e.g., due to severe cognitive impairment or communication problems)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of 207 geriatric patients aged 65 years and older who were admitted to the emergency department with a diagnosis of acute coronary syndrome (ACS)
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | Within 30 days after emergency department admission
  Occurrence of major adverse cardiac events (MACE) including STEMI, NSTEMI, unstable angina, or cardiovascular mortality.

SECONDARY OUTCOMES:
Physical Activity Score (IPAQ-SF) | At baseline (hospital admission, emergency department evaluation)
  Physical activity level measured using the International Physical Activity Questionnaire Short Form (IPAQ-SF). Score range: 0 to 1920 MET-minutes/week. Higher scores indicate greater levels of physical activity.
TIMI Risk Score | At baseline (emergency department evaluation)
  Thrombolysis in Myocardial Infarction (TIMI) Risk Score. Risk stratification assessed using the TIMI Risk Score, which is based on clinical history, electrocardiogram findings, troponin levels, and cardiovascular risk factors. Score range: 0 to 7. Higher scores indicate greater risk and worse prognosis.
HEART Risk Score | At baseline (emergency department evaluation)
  HEART Risk Score (History, Electrocardiogram, Age, Risk factors, Troponin). Risk stratification assessed using the HEART Risk Score, which is based on patient history, electrocardiogram findings, age, cardiovascular risk factors, and troponin levels. Score range: 0 to 10. Higher scores indicate increased risk of major adverse cardiac events (worse prognosis).
SVEAT Risk Score | At baseline (emergency department evaluation)
  SVEAT Risk Score (Symptoms, Vascular disease, Electrocardiogram, Age, Troponin). Risk stratification assessed using the SVEAT Risk Score, based on symptoms, history of vascular disease, electrocardiogram findings, age, and troponin levels. Score range: 0 to 10. Higher scores indicate increased cardiovascular risk and worse prognosis.
All-cause Mortality | Within 30 days after admission
  Death from any cause among study participants after acute coronary syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Balıkesir University Faculty of Sport Sciences / Department of Coaching Education, Balıkesir, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is retrospective and based on hospital records, and data sharing is restricted due to patient privacy and ethical considerations.